CLINICAL TRIAL: NCT02108054
Title: Behavioral and Functional Task Development, Implementation, and Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 140066; 14-AA-0066
Record Dates: First submitted 2014-04-08; First posted 2014-04-09 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2025-12-03

CONDITIONS: Alcohol Dependence; Alcohol Drinking; Alcoholism; Alcohol Use Disorder; Addiction
Keywords: fMRI; Alcoholism; Phenotype; Imaging; EEG; Psychophysiology; Near Infrared
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Behavior, Addictive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): People with alcohol use disorder
  Interventions: Device: 7T MRI
- 2 (Experimental): People without alcohol use disorder
  Interventions: Device: 7T MRI

INTERVENTIONS:
Device: 7T MRI — Modifying, refining, and verifying the feasibility and applicability of tasks for functional magnetic resonance imaging (fMRI) to measure intended concomitant brain activation

SUMMARY:
Background:

- Scientists know that alcohol use disorders affect brain structure. They want to know more about the effects of alcohol use disorders on a person s behavior. They want to develop tasks that can be done inside a scanner that can help them better understand these effects in later studies.

Objective:

- To develop tasks that investigate a person s behavior that can be used in later studies.

Eligibility:

* Inpatient participants of another study. They must be physically healthy right-handed adults 18-60 years old.
* Healthy right-handed volunteers 18-65 years old.

Design:

* Participants will be screened with medical history and physical exam. They will have an EKG to record heart activity. They will give blood and urine samples and have a psychiatric interview.
* Participants will have between one and three visits.
* Participants will be asked about their alcohol drinking to see if they have an alcohol use disorder.
* Participants will complete one of three simple computerized tasks either inside the magnetic resonance imagining (MRI) scanner or outside of it.
* The MRI scanner takes pictures of the brain. The scanner is a metal cylinder. Participants lie on a table that can slide in and out of the cylinder. They will be in the scanner for about 60 minutes. They may have to lie still for up to 20 minutes. The scanner makes loud knocking noises, but they will get earplugs.

DETAILED DESCRIPTION:
Objective:

The purpose of this protocol is three-fold: 1) to develop tasks examining various cognitive, motivational, and decision-making behaviors outside the scanner; 2) to modify, refine, and verify the feasibility and applicability of tasks for functional magnetic resonance imaging (fMRI) to measure intended concomitant brain activation; and 3) to examine equivalent or surrogate signals using other devices such as electroencephalograph (EEG) and functional near infrared spectrometer (fNIRS) when the MR contraindication(s) are present in the participant.

Study population:

Healthy volunteers without an alcohol use disorder, and inpatient participants with alcohol dependence as determined by the DSM-IV-TR or at least Moderate Alcohol Use Disorder as determined by DSM-5.

Design:

The participants will pilot one or both aspects of this study depending on whether the task is de novo or a modification to previously verified or published task.

Outcome measures:

The outcome is to develop and examine tasks that reliably measure specific cognitive, motivational and decision-making behaviors and invoke associated brain systems and functions in our targeted subject populations.

ELIGIBILITY:
* INCLUSION CRITERIA:
* between 18-65 years of age. The PI or designated AI will determine if any of the exclusion criteria listed below applies*.

EXCLUSION CRITERIA:

* Are not cleared on a neuromotor examination
* Are currently receiving psychotropic medication
* Inpatients only: Currently experiencing symptoms of withdrawal from alcohol (As determined by the most recent measurement within the

past 30 days CIWA score > 8).

-MRI Exclusion Criteria:

* Presence of ferromagnetic objects in the body including implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metallic fragments in the eye that welders and other metal workers may have;
* Are pregnant, as determined by a negative pregnancy test
* Left handed
* Claustrophobia.

  * To minimize discomfort and undue burden on the participants, unless available from phone screening, pre-screening, or other NIAAA studies such as 14-AA-0080, 14-AA-0181, we collect the above information as part of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
outcome is to develop and examine tasks that reliably measure specific cognitive, motivational and decision-making behaviors | ONGOING
  Tasks that are suitable for fMRI studies and other clinical research measurements

CONTACTS AND LOCATIONS:
Overall Officials: Paule V Joseph, C.R.N.P., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study is designed to determine and modify tasks to induce and affect various behavioral, psychophysiological and neural responses. Therefore, it appears that in order to make such data available they should be collected in future hypothesis driven studies that utilize the tasks developed under this protocol.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-AA-0066.html